CLINICAL TRIAL: NCT04077229
Title: Piloting Text Messages to Promote Positive Affect and Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Associate Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001472
Record Dates: First submitted 2019-08-28; First posted 2019-09-04 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS; Text Message; Positive Psychology; Health Behavior
MeSH Terms: conditions — Acute Coronary Syndrome; Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): A total of 28 intervention text messages (1/day for 4 weeks) will be sent to participants following the baseline self-report assessment. After each message is sent, participants will receive a second text message asking them to rate the utility of the message. Following the 4-week intervention, participants will complete the same self-report assessments as in the baseline assessment (via phone) and will provide feedback about the program. Finally, 4 weeks later (at 8 weeks), participants will repeat the self-report questionnaires by phone.
  Interventions: Behavioral: Intervention arm: Text Message Intervention

INTERVENTIONS:
Behavioral: Intervention arm: Text Message Intervention — Participants will receive a combination of messages promoting both psychological well-being and education /support around health behavior adherence, such as physical activity or diet. In the first part of the study, participants will receive 28 fixed text messages that alternate between physical activity and PP (Positive Psychology) messages. In the second part of the study, participants will first receive a set of 14 pre-selected daily messages that contain a broad range of attributes to allow sufficient participant feedback to clearly identify preferences. After the first 14 messages, new messages will be selected based on the prior preferences of participants.

SUMMARY:
The focus of the study is to assess the feasibility and acceptability of a pilot one-arm project delivering text messages related to positive psychology (PP) activities (e.g., recalling positive events) and health behavior text messages (e.g. having a heart-healthy diet, becoming more physically active). The messages will be sent for 4 weeks among patients with a prior acute coronary syndrome (ACS).

DETAILED DESCRIPTION:
This is a single-arm study of text messaging in post-ACS patients. The convenience sample for this pilot study will be enrolled from two sources: (a) participants prospectively enrolled from inpatient cardiac units at MGH admitted for an ACS, and (b) participants in prior post-ACS studies performed with the investigators' team.

A total of 28 intervention text messages (1/day for 4 weeks) will be sent to participants following the baseline assessment. After each message is sent, participants will receive a second text message asking them to rate the utility of the message, and this rating will be used by a machine learning algorithm to select subsequent messages. This will ensure that, over time, participants will receive messages that they are more likely to find useful.

In the first part of the study, participants will receive 28 fixed text messages that alternate between physical activity and positive psychology messages. In the second part of the study, participants will receive 14 fixed text messages that range in topics from positive psychology to physical activity, diet, and medication adherence. In the second part of the study, participants will first receive a set of 14 pre-selected daily messages that contain a broad range of attributes to allow sufficient participant feedback to clearly identify preferences. After the first 14 messages, new messages will be selected based on the prior preferences of participants.

The messages will be sent using the Twilio texting program used by REDCap, which also uses Amazon Web Services. Twilio allows software developers to programmatically make and receive phone calls and send and receive text messages using its web service. The investigators have purchased a Twilio account to allow messages to come from an anonymous phone number rather than the phone of a study staff member.

ELIGIBILITY:
Inclusion Criteria:

1. Prior acute coronary syndrome.

   Acute myocardial infarction (MI):
   * Elevation of cardiac biomarkers (cardiac troponin T) in addition to one or more of the following:
   * symptoms of ischemia (e.g., acute chest pain)
   * ischemic changes on electrocardiogram
   * imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

   Unstable angina (UA):
   * crescendo angina
   * new onset (within 1 month) angina with minimal exertion
   * angina with minimal exertion or at rest.
2. Ability to receive text messages via cellular phone.

Exclusion Criteria:

* A periprocedural ACS
* Terminal illness
* An unrelated condition limiting physical activity
* An inability to communicate in English, or
* cognitive disorder assessed by 6-item cognitive screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Percentage of text messages successfully delivered to participants | 4 weeks
  Feasibility will be measured by calculating the percentage of text messages successfully delivered to participants.
Participant burden | 4 weeks
  Mean ratings of the intervention's burden, as reported by participants on a 0-10 Likert-type scale (0= not burdensome at all; 10= extremely burdensome).
Self-reported utility of the intervention | 4 weeks
  Mean ratings of the intervention's utility, as reported by participants on a 0-10 Likert-type scale (0= not helpful at all; 10= extremely helpful).

SECONDARY OUTCOMES:
Change in Positive Affect at 4 weeks | Change in positive affect from baseline to 4 weeks
  Pre-post changes in level of positive affect on a 0-10 Likert scale (0=not happy at all, 10-extremely happy). Higher values represent a better outcome.
Change in Positive Affect at 8 weeks | Change in positive affect from baseline to 8 weeks
  Pre-post changes in level of positive affect on a 0-10 Likert scale (0=not happy at all, 10-extremely happy). Higher values represent a better outcome.
Change in Optimism at 4 weeks | Change in optimism from baseline to 4 weeks
  Pre-post changes in level of optimism on a 0-10 Likert scale (0=not optimistic at all, 10-extremely optimistic). Higher values represent a better outcome.
Change in Optimism at 8 weeks | Change in optimism from baseline to 8 weeks
  Pre-post changes in level of optimism on a 0-10 Likert scale (0=not optimistic at all, 10-extremely optimistic). Higher values represent a better outcome.
Change in Determination at 4 weeks | Change in determination from baseline to 4 weeks
  Pre-post changes in level of determination on a 0-10 Likert scale (0=not determined at all, 10= extremely determined). Higher values represent a better outcome.
Change in Determination at 8 weeks | Change in determination from baseline to 8 weeks
  Pre-post changes in level of determination on a 0-10 Likert scale (0=not determined at all, 10= extremely determined). Higher values represent a better outcome.
Change in Depression at 4 weeks | Change in depression from baseline to 4 weeks
  Pre-post changes in level of depression on a 0-10 Likert scale (0=not depressed at all, 10= extremely depressed). Higher values represent a better outcome.
Change in Depression at 8 weeks | Change in depression from baseline to 8 weeks
  Pre-post changes in level of depression on a 0-10 Likert scale (0=not depressed at all, 10= extremely depressed). Higher values represent a better outcome.
Change in Anxiety at 4 weeks | Change in anxiety from baseline to 4 weeks
  Pre-post changes in level of anxiety on a 0-10 Likert scale (0=not anxious at all, 10= extremely anxious). Higher values represent a better outcome.
Change in Anxiety at 8 weeks | Change in anxiety from baseline to 8 weeks
  Pre-post changes in level of anxiety on a 0-10 Likert scale (0=not anxious at all, 10= extremely anxious). Higher values represent a better outcome.
Change in Self-reported physical activity at 4 weeks | Change in self-reported physical activity from baseline to 4 weeks
  Pre-post changes in level of physical activity. Participants will complete a two-item assessment for physical activity that has been validated and used in thousands of patients in the Kaiser Permanente system. We will record completion of moderate activity in number of minutes of activity/week. The items are:
  In the past 4 weeks, how many days/week did you engage in moderate or greater physical activity? On those days, how many minutes do you engage in activity at this level? These two measures are multiplied to arrive at the average min/week of moderate or greater physical activity.
Change in Self-reported physical activity at 8 weeks | Change in self-reported physical activity from baseline to 8 weeks
  Pre-post changes in level of physical activity. Participants will complete a two-item assessment for physical activity that has been validated and used in thousands of patients in the Kaiser Permanente system. We will record completion of moderate activity in number of minutes of activity/week. The items are:
  In the past 4 weeks, how many days/week did you engage in moderate or greater physical activity? On those days, how many minutes do you engage in activity at this level? These two measures are multiplied to arrive at the average min/week of moderate or greater physical activity.
Change in Self-reported dietary adherence at 4 weeks | Change in dietary adherence from baseline to 4 weeks
  Pre-post changes in level of self-reported dietary adherence. Participants will be asked a single item about self-reported dietary adherence, adapted from the Medical Outcomes Study Specific Adherence Scale. "In the last month, how often have you followed a low-fat, low-salt, or other diet as prescribed by your treatment team?" Choices will include "None of the time (1)," "A little of the time (2)," "Some of the time (3)," "A good bit of the time (4)," "most of the time (5)," and "all of the time (6)." Higher values represent a better outcome.
Change in Self-reported dietary adherence at 8 weeks | Change in dietary adherence from baseline to 8 weeks
  Pre-post changes in level of self-reported dietary adherence. Participants will be asked a single item about self-reported dietary adherence, adapted from the Medical Outcomes Study Specific Adherence Scale. "In the last month, how often have you followed a low-fat, low-salt, or other diet as prescribed by your treatment team?" Choices will include "None of the time (1)," "A little of the time (2)," "Some of the time (3)," "A good bit of the time (4)," "most of the time (5)," and "all of the time (6)." Higher values represent a better outcome.
Change in Self-reported health/function at 4 weeks | Change in self-reported health/function from baseline to 4 weeks
  Participants will be asked a single item about self-reported health: "In general, how would you rate your health today" with the possible choices being "very good" (1), "good" (2), "moderate" (3), "bad" (4) or "very bad" (5). This scale is a robust predictor of mortality and correlates strongly with other objective health indicators. Lower values represent a better outcome.
Change in Self-reported health/function at 8 weeks | Change in self-reported health/function from baseline to 8 weeks
  Participants will be asked a single item about self-reported health: "In general, how would you rate your health today" with the possible choices being "very good" (1), "good" (2), "moderate" (3), "bad" (4) or "very bad" (5). This scale is a robust predictor of mortality and correlates strongly with other objective health indicators. Lower values represent a better outcome.
Change in self-reported physical function at 4 weeks | Change in self-reported physical function from baseline to 4 weeks
  This will be assessed with the Duke Activity Status Index (DASI). The DASI contains 12 items that inquire about activities of daily living (e.g., bathing), basic physical activity (e.g., walking, climbing stairs), and more strenuous physical function (e.g., vigorous sports) to gauge overall functional capacity. Higher values represent a better outcome (range 0-58.2).
Change in self-reported physical function at 8 weeks | Change in self-reported physical function from baseline to 8 weeks
  This will be assessed with the Duke Activity Status Index (DASI). The DASI contains 12 items that inquire about activities of daily living (e.g., bathing), basic physical activity (e.g., walking, climbing stairs), and more strenuous physical function (e.g., vigorous sports) to gauge overall functional capacity. Higher values represent a better outcome (range 0-58.2).

CONTACTS AND LOCATIONS:
Locations (1):
- Jeff Huffman, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT04077229/Prot_SAP_000.pdf